CLINICAL TRIAL: NCT02225002
Title: Phase 1, Open-Label, Dose-Escalation Study of CP-870,893 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: UPCC 10903
Record Dates: First submitted 2014-08-22; First posted 2014-08-25 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Advanced Solid Tumors
Keywords: relapsed; refractory to standard therapy; no effective therapy exists
MeSH Terms: conditions — Recurrence | interventions — selicrelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CP-870,893

SUMMARY:
CD40, a member of the Tumor Necrosis Factor receptor superfamily, is expressed on many tumor types, including melanoma, prostate, colon, breast, renal, pancreatic, and nonsmall cell lung cancers. In preclinical models, activation of CD40 results in increased antigen presentation and induction of apoptosis. CD40 is also expressed on antigen presenting cells (APCs) (B cells, dendritic cells, monocytes) and is a key regulator of both cellular and humoral immune responses. Activation of CD40 by CP-870,893, an agonistic anti-CD40 monoclonal antibody, enhances host immune responses and abrogates the growth of tumors independently of the expression of CD40 on tumor cells. Therefore, it is hypothesized that therapeutic intervention with CP-870,893 may be beneficial to a large number of cancer patients either through an immunomodulatory effect or through a direct effect on CD40-positive tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years old with advanced solid tumors relapsed or refractory to standard therapy or for whom no effective therapy exists;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1;
* Adequate bone marrow function documented within 2 weeks prior to treatment, defined as:
* White blood cell (WBC) count >3000 cells/μL without growth factor support;
* Absolute neutrophil count (ANC) ≥1500/μL without growth factor support;
* Platelets >100,000/μL without growth factor support; and
* Hemoglobin ≥10 g/dL;
* D-dimer WNL;
* Adequate renal and hepatic function documented within 2 weeks prior to treatment, defined as:
* Total bilirubin <1.5 times the upper limit of normal (ULN);
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) <2.5 × ULN;
* Creatinine clearance (CLcr, measured or calculated) >80 mL/min; and
* Life expectancy of at least 12 weeks;
* Fully recovered from the acute effects of prior cancer therapy: 4 weeks for chemotherapy (8 weeks for mitomycin C or nitrosoureas), 10 days for prior palliative radiation therapy or hormonal therapy, and 4 weeks for prior immunotherapy or other biologic therapy; and
* Signed written informed consent.

Exclusion Criteria:

* Previously treated with any other agent that targets CD40;
* Concurrent treatment with any anticancer agent;
* History of autoimmune disorder, including pemphigus vulgaris, systemic mastocytosis, systemic lupus erythamatosus, dermatomyositis/polymyositis, rheumatoid arthritis, systemic sclerosis, Sjörgen's syndrome, vasculitis/arteritis, Behcet's syndrome, inflammatory boweldisease, autoimmune thyroiditis, multiple sclerosis, or other chronic inflammatory disease;
* Treatment with any other investigational therapy within 4 weeks prior to baseline;
* History (within the previous year) of congestive heart failure, stroke, or myocardial infarction;
* Patients with known hereditary or acquired coagulopathies (eg. hemophilia, von Willebrand's disease, cancer-associated DIC, abnormal D-dimer);
* Patients with known brain metastases. Patients with clinical evidence suggestive of new brain metastases prior to enrollment are excluded if brain metastases have not been ruled out via CT or MRI. Patients with previously diagnosed brain metastases are eligible if they have completed their CNS treatment and have recovered from the acute effects of radiation therapy or surgery prior to the start of study medication, have discontinued corticosteroid treatment for these metastases for at least 4 weeks, and are neurologically stable;
* Patients having reproductive potential who are not using an effective method of birth control or who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test during baseline;
* Known sensitivity to immunomodulating agents or monoclonal antibodies;
* Alcohol abuse or illicit drug use within 12 months of enrollment;
* History of serum creatinine ≥2 mg/dL for any duration and for any reason;
* Patients, other than menstruating females, with urine dipstick 1+ or more positive for blood or 2+ or more positive for protein;
* Patients with clinically significant presence of granular or cellular casts in centrifuged urine sediment;
* Patients with renal carcinoma or renal metastases;
* Patients that have had a partial or complete nephrectomy;
* Patients requiring dialysis (peritoneal or hemodialysis);
* Prior treatment with Amphotericin B or cisplatin;
* Patients with history of insulin-dependent diabetes for greater than 5 years;
* Concomitant treatment with systemic high dose corticosteroids or treatment with systemic corticosteroids within 4 weeks of baseline;
* Concomitant treatment with anticoagulants, such as coumadin or heparin, except to maintain patency of in-dwelling catheters;
* Prior allergic reactions attributed to compounds of similar chemical or biologic composition to study drug (eg, rituximab or immunoglobulin G);
* Ongoing or active infection;
* Required the use of systemic antibiotics or antifungals for ongoing or recurrent infections.

Topical use of antibiotics or antifungals is allowed;

* Other uncontrolled concurrent illness that would preclude study participation; or
* Psychiatric illness or social situation that would preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vonderheide, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States